CLINICAL TRIAL: NCT03026920
Title: Different Surgical Methods for Pelvic or Acetabular Fracture of Old Man
Brief Title: Pelvic and Acetabular Fracture in Old People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZY2015
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-01

CONDITIONS: Fracture Dislocation
Keywords: Fracture; outcome; pelvic; acetabular
MeSH Terms: conditions — Fracture Dislocation; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clinical outcome (Experimental): Less invasive method was applied to pelvic or acetabular fracture of old people. Thus, the clinical outcome of Pelvic or acetabular fractures in old man was assessed.
  Interventions: Procedure: less invasive method

INTERVENTIONS:
Procedure: less invasive method — The less invasive surgical method was conducted in this study. Then, the clinical results were compared with the patients treated using traditional methods to assess the less invasive method.

SUMMARY:
It was reported that satisfactory postoperative outcome was difficult to obtain for the pelvic or acetabular fracture in old people. The less invasive surgical method was conducted in this study. Then, the clinical results were compared with the patients treated using traditional methods to assess the less invasive method.

DETAILED DESCRIPTION:
Pelvic or acetabular fractures were caused by high energy trauma, which may lead to poor prognosis for the old. The patients over 60 years were included in this study. The surgical procedure was conducted in two weeks. The less invasive methods involved Stoppa approach and novel plate. The data including surgical time, blood loss and results of follow-up were recorded. The clinical results were compared with the patients treated using traditional methods. Thus, the clinical outcome of Pelvic or acetabular fractures in old man was assessed.

ELIGIBILITY:
Inclusion Criteria:

Over 60 years old Fracture involving pelvis or acetabulum Operation was conducted within 14 days Sign the consent form

Exclusion Criteria:

Presented with a pathologic acetabular fracture Refused to participate Follow-up insufficient 12 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
fracture union time | 4 months
  how long the fracture line disappeared postoperatively in radiograph

SECONDARY OUTCOMES:
complication | 12 months
  wound infection, iatrogenic injury of vessels and nerves, nonunion

CONTACTS AND LOCATIONS:
Overall Officials: Ruipeng Zhang, M.D, Principal Investigator — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No